CLINICAL TRIAL: NCT03787680
Title: A Multi-Center Phase II Study Testing the Activity of Olaparib and AZD6738 (ATR Inhibitor) in Metastatic Castration-Resistant Prostate Cancer
Brief Title: Targeting Resistant Prostate Cancer With ATR and PARP Inhibition (TRAP Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.108; HUM00152799 (Other: University of Michigan)
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; ceralasertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (DRPro) (Experimental): Patients with metastatic castration-resistant prostate cancer (mCRPC) who are DNA repair proficient (DRPro).
  Interventions: Drug: Olaparib; Drug: AZD6738
- Cohort 2 (DRDef) (Experimental): Patients with metastatic castration-resistant prostate cancer (mCRPC) who are DNA repair deficient (DRDef).
  Interventions: Drug: Olaparib; Drug: AZD6738

INTERVENTIONS:
Drug: Olaparib — 300 mg by mouth twice a day for days 1-28 of a 28-day cycle.
  Other Names: AZD2281; ceralasertib
Drug: AZD6738 — 160 mg by mouth daily for days 1-7 of a 28-day cycle.

SUMMARY:
The purpose of this study is to test the effectiveness (how well the drugs work), safety, and tolerability of the investigational drug combination of olaparib and AZD6738 for all patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male ages 18 years and older at time of signing the informed consent form
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 within 42 days prior to registration
4. Histologic or cytologic proof of prostate adenocarcinoma (excluding small-cell or neuroendocrine pathologies)
5. Metastatic prostate cancer on CT, MRI or Bone scan
6. Must have disease progression (while testosterone level is under 50 ng/dl) on prior therapy prior to study entry defined as one (or more) of the following:

   1. PSA progression defined as continuously rising PSA values measured a minimum of 1 week apart with a minimal starting value of 1.0 ng/mL
   2. Progression of bidimensionally measurable soft tissue or nodal metastasis by CT or MRI based on RECIST, v1.1
7. Prior treatment with at least one of the following:

   1. One line of therapy in mCRPC
   2. Second generation anti-androgen (e.g. abiraterone, enzalutamide or apalutamide) within the hormone-sensitive phase of disease AND progression occurs while on therapy
8. Patients must be withdrawn from prior therapy for ≥3 weeks (patients may remain on prior prednisone up to 10 mg total daily exposure at provider's discretion) at planned time of treatment start.
9. Agree to undergo a biopsy of at least one metastatic site (if feasible) to determine DNA repair status, unless prior metastatic tissue underwent next-generation sequencing in a CLIA certified lab or known germline loss of BRCA1, BRCA2 or ATM. If no site is reachable, or first biopsy insufficient/unsuccessful, circulating tumor DNA may be obtained.
10. Treated with continuous androgen deprivation therapy (either surgical castration or LHRH agonist/antagonist) with documented castrate level of serum testosterone (<50 ng/dL). A stable dose of bisphosphonate or denosumab for bone metastases should be continued as long as started at least 5 days prior to C1D1 planned start day.
11. At the time of planned treatment start (C1D1), at least 21 or more days will have elapsed from palliative radiation (with the exception of radiation to >30% of bone marrow or with a wide field of radiation, this requires 28 or more days).
12. Patient must have normal organ and bone marrow function measured within 42 days prior to registration as defined below

    1. Hemoglobin ≥10 g/dL (with no blood transfusion or erythropoietin use within the past 42 days)
    2. Absolute neutrophil count ≥1.5x109/L
    3. Platelet count ≥100x109/L (with no platelet transfusions within last 42 days)
    4. Total bilirubin <1.5x ULN (unless the patient has documented Gilbert's disease and <2.0x ULN should be used)
    5. AST or ALT ≤ 2.5x ULN, unless liver metastases are present in which case they cannot be ≥5x ULN
    6. Glomerular filtration rate (GFR) ≥51 mL/min, as assessed using the Cockcroft- Gault equation
13. Estimated life expectancy ≥16 weeks
14. Male patients who are sexually active must be willing to use barrier contraception for the duration of the study and for 1 week after the last study drug administration, with all sexual partners. Male patients must use a condom during treatment and for 6 months after the last dose of study drug(s) when having sexual intercourse with a pregnant woman or with a woman of childbearing potential and must not donate sperm for 6 months after the last dose of study drug. Female partners of male patients should also use a highly effective form of contraception (per protocol) for 6 months after the last dose of study drug(s) if they are of childbearing potential. True abstinence is an acceptable form of contraception and must be documented as such.
15. Patient is willing and able to comply with the protocol for the duration of the study, including undergoing biopsy (if warranted), treatment, scheduled visits and examinations

Exclusion Criteria:

1. A diagnosis of ataxia telangiectasia
2. Prior treatment with a PARP inhibitor (e.g. olaparib, veliparib, niraparib, rucaparib), AZD6738 or other DNA-damage response agents (e.g. cisplatin or carboplatin)
3. Cytotoxic chemotherapy, first- or second-generation antiandrogen or CYP17 inhibitors are not permitted within 21 days or 5 half-lives of registration (whichever is longest) of planned treatment start. For clarity, enzalutamide requires 5 weeks washout.
4. Major surgery < 2 weeks prior to enrolment; patients must have recovered from any effects of major surgery
5. Persistent toxicities (≥CTCAE Grade 2) caused by previous cancer therapy, besides Grade 2 alopecia and Grade 2 neuropathy (these are allowed).
6. Patients with current or prior MDS/AML or with features suggestive of MDS/AML
7. Any other malignancy which has been active or treated within the past 3 years, with the exception of non-melanomatous skin cancer, or Ta bladder cancer
8. Patients with active brain metastases are excluded because of unknown penetration into the CNS. A confirmatory scan for asymptomatic patients is not required. Patients with a history of treated central nervous system (CNS) metastases are eligible provided they meet all of the following criteria: disease outside the CNS is present, no clinical evidence of progression since completion of CNS-directed therapy, minimum 3 weeks between completion of radiotherapy and registration and recovery from significant (Grade ≥ 3) acute toxicity with no ongoing requirement for >10 mg of prednisone per day or an equivalent dose of other corticosteroid. If a patient must remain on steroids, they must have started the steady dose at least 28 days prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days prior to study treatment.
9. Any of the following cardiac disease currently or within the last 6 months:

   1. Unstable angina pectoris
   2. Congestive heart failure (by New York Heart Association ≥ Class 2) or known reduced LVEF < 55%
   3. Acute myocardial infarction
   4. Conduction abnormality not controlled with pacemaker or medication (e.g. complete left bundle branch block or third-degree heart block)
   5. Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
   6. Uncontrolled hypertension (Grade 2 or above) requiring urgent (for example, adjusting medications within 24 hours) clinical intervention
   7. Patients at risk of brain perfusion problems, e.g. TIAs or history of pre- syncope or syncopal episodes unexplained by reversible causes
10. Mean resting corrected QT interval >450, obtained from 3 ECGs 2-5 minutes apart using the Fredericia formula. Absence of any factors that increase the risk of QTc prolongation or risk of arrhythmic such as congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 year of age. Patients with relative hypotension (<90/60 mmHg) or previously known clinically relevant orthostatic hypotension defined as a postural hypotension ≥20 mmHg
11. Concomitant use of known potent or moderate cytochrome P (CYP) 3A inhibitors (e.g. itraconazole, ciprofloxacin, diltiazem) require 2-week washout prior to planned C1D1. Concomitant use of strong or moderate CYP3A inducers (e.g. phenobarbital, enzalutamide, modafinil require 5-week washout for enzalutamide or phenobarbital and 3 week washout for all others, per protocol.
12. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases that places the patient at unacceptable risk of toxicity or non-compliance. Examples include, but are not limited to, active bleeding diatheses, renal transplant, uncontrolled major seizure disorder, severe COPD, superior vena cava syndrome, extensive bilateral lung disease on High Resolution CT scan, severe Parkinson's disease, active inflammatory bowel disease, psychiatric condition, immunocompromised patients or active infection including any patient known to have hepatitis B, hepatitis C and human immunodeficiency virus (HIV) or requiring systemic antibiotics, antifungals or antiviral drugs. Screening for chronic conditions is not required
13. A known hypersensitivity to olaparib, AZD6738 or any excipient of the product or any contraindication to the combination anti-cancer agent as per local prescribing information
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with the absorption of the study medication, refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of AZD6738
15. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
16. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.12)
17. Involvement in the planning and/or conduct of the study
18. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
19. Previous enrolment in the present study.
20. Has received a live vaccination with 2 weeks of enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2028-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zachery Reichert, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (DRPro) | Cohort 2 (DRDef)
Started | 37 | 12
Completed | 26 | 5
Not Completed | 11 | 7
Not completed — Physician Decision | 2 | 3
Not completed — Adverse Event | 7 | 3
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (DRPro) | Cohort 2 (DRDef) | Total
Number analyzed (Participants) | 37 | 12 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 27 | 8 | 35
Age, Continuous [Mean (Full Range); unit: years] | 70.2 [54 to 88] | 67.9 [54 to 81] | 69 [54 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 12 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 34 | 10 | 44
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 28 | 12 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 37 | 12 | 49

OUTCOME MEASURES:

1. Primary Outcome: Rate of Response (Complete Response [CR] or Partial Response [PR]) in DNA Repair Proficient (DRPro) Patients
Description: Evaluated per radiographic response according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or by Prostate Specific Antigen (PSA) (≥50% decline).
Time Frame: Up to 30 days after study completion (an average of 1 year)
Population: this endpoint only applies to DRPro patients
Measure: Number; unit: percentage of patients
Arm/Group | Cohort 1 (DRPro) | Cohort 2 (DRDef)
Number analyzed (Participants) | 37 | 0
percentage of patients | 11.4 |

2. Secondary Outcome: Rate of Response (Complete Response [CR] or Partial Response [PR]) in DNA Repair Deficient (DRDef) Patients
Description: Evaluated per radiographic response according to RECIST v1.1 or PSA (≥50% decline).
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival (PFS) in DRPro Patients
Description: Duration of time from start of treatment to time of progression (based only on radiographic progression or clinical decline/death).
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free Survival (PFS) in DRDef Patients
Description: as for outcome 3
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

5. Secondary Outcome: Radiographic Response Rate in DRPro Patients
Description: Evaluated according to RECIST v1.1.
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

6. Secondary Outcome: Radiographic Response Rate in DRDef Patients
Description: Evaluated according to RECIST v1.1.
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

7. Secondary Outcome: PSA Progression-free Survival in DRPro Patients
Description: Composite of survival and duration of PSA control as defined by time from start of therapy to first PSA increase ≥ 25% and ≥2 ng/ml above the nadir and confirmed by a second value at or beyond 4 weeks later.
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

8. Secondary Outcome: PSA Progression-free Survival in DRDef Patients
Description: as for outcome 7
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

9. Secondary Outcome: PSA Response Rate in DRPro Patients
Description: Rate of achieving PSA response rate of ≤ 0.2 ng/ml, 50% decline, or 90% decline from entry PSA and confirmed 4 weeks later
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

10. Secondary Outcome: PSA Response Rate in DRDef Patients
Description: as for outcome 9
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

11. Secondary Outcome: Duration of Combined Radiographic and PSA Response in DRPro Patients
Description: Time from first documented response (RECIST v1.1 CR/PR or PSA decline ≥50%) until death, recurrent or progressive disease (based on RECIST v1.1) or first PSA increase ≥ 25% and ≥2 ng/ml above the PSA nadir.
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

12. Secondary Outcome: Duration of Combined Radiographic and PSA Response in DRDef Patients
Description: as for outcome 11
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

13. Secondary Outcome: Adverse Events
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: Up to 30 days after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

14. Secondary Outcome: Incidence of Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML) and New Primary Malignancy
Time Frame: Up to 5 years after study completion (an average of 1 year for study completion)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 3.5 year period.
Arm/Group | Cohort 1 (DRPro) | Cohort 2 (DRDef)
All-Cause Mortality (participants affected / at risk) | 22/37 | 7/12
Serious Adverse Events (participants affected / at risk) | 2/37 | 4/12
Other Adverse Events (participants affected / at risk) | 35/37 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (DRPro) (N=37) | Cohort 2 (DRDef) (N=12)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Erroneous administration
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — submandibular abscess
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (DRPro) (N=37) | Cohort 2 (DRDef) (N=12)
Anemia (Blood and lymphatic system disorders) | 24 (69) | 8 (23)
Anorexia (Metabolism and nutrition disorders) | 7 (10) | 3 (3)
Creatinine increased (Investigations) | 5 (8) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (3)
Fatigue (General disorders) | 18 (30) | 6 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (12) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (7) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (25) | 6 (10)
Platelet count decreased (Investigations) | 5 (6) | 1 (1)
White blood cell decreased (Investigations) | 7 (17) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT03787680/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03787680/ICF_001.pdf